CLINICAL TRIAL: NCT00354705
Title: Prognostic Molecular and Environmental Factors in High-Risk Stage II and Stage III Colon Cancer Patients
Brief Title: Prognostic Molecular and Environmental Factors in High-Risk Colon Cancer Patients
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 2005-0383
Record Dates: First submitted 2006-07-18; First posted 2006-07-20 (Estimated); Last update posted 2019-05-10 (Actual); Status verified 2019-05

CONDITIONS: Colon Cancer
Keywords: Colon Cancer; Adenocarcinoma of the Colon; Cancer Recurrence; Survey; Chemotherapy; Surgery
MeSH Terms: conditions — Colonic Neoplasms | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — 20 ml of blood for genomic analysis collected at baseline, at completion of adjuvant chemotherapy ( <28 days after its completion) if applicable, at each subsequent surveillance visit (every 3 months after discontinuation of adjuvant chemotherapy, continuing for 2 years), and at time of disease recurrence, if applicable.
  20 ml of blood for proteomic analysis studies collected at baseline, at completion of adjuvant chemotherapy, if applicable ( <28 days after its completion), and at time of disease recurrence, if applicable.
  Tissue (0.2gm of tissue) from primary resection obtained at time of study enrollment. A tissue sample (0.2gm of tissue) also obtained, if possible, from patients that require surgical intervention at M.D. Anderson Cancer Center, for recurrent disease.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Colon Cancer Patients: Patients with colon cancer recently removed by surgery.
  Interventions: Behavioral: Questionnaire

INTERVENTIONS:
Behavioral: Questionnaire — Two questionnaires taking 30 minutes to complete.
  Other Names: Survey

SUMMARY:
The goal of this research study is to identify biologic and lifestyle factors that may increase a person's risk of developing a recurrence (return) of colon cancer.

DETAILED DESCRIPTION:
Treatment with drugs (chemotherapy) and frequent evaluations by a doctor are standard practice to help prevent colon cancer from recurring after surgery. Despite these measures, the cancer does recur in a significant number of people, usually within the first 2-3 years from diagnosis.

In this study, researchers hope to identify genetic and environmental factors that may contribute to a person developing recurrent colon cancer. To help identify these factors, blood and tissue samples will be studied. You also will be asked to provide information about your background, lifestyle, and eating habits.

Participants able to take part in this study have had all of their known colon cancer removed by surgery and have agreed to receive chemotherapy to help prevent the cancer from recurring. Before you take part in this study, your medical information will be reviewed, and a performance status evaluation (how well you perform everyday activities) will be done. This will help the doctor decide if you are eligible to take part in the study.

If you are found to be eligible and you agree to take part in the study, you will be asked to fill out 2 questionnaires. One questionnaire asks about your background (age, education, etc.), work history, any exposure to toxic substances, medical history, smoking and alcohol history, family history of cancer, and your level of physical activity. The second questionnaire contains questions about what types of foods you eat, how often you eat them, whether you take vitamins and if so, what type(s). It will take about 30 minutes to fill out both of these questionnaires.

If your surgery to remove your colon cancer was not performed at MD Anderson, you will not be asked to participate in the tissue portion of this study described below but you will be asked to participate in the blood sample analysis and the study evaluations and questionnaire portion of this study every 3 months for a maximum of 2 years (starting from the beginning of the follow-up period, once all treatment is complete) or until your disease returns, which ever occurs first.

If your surgery was performed at MD Anderson Cancer Center, the samples of your cancer tissue will be analyzed, looking for any biologic factors related to colon cancer. Blood samples (about 4 teaspoons) for gene analysis (looking for any biologic factors associated with colon cancer) will also be collected.

Once follow-up begins, you will have study evaluations at MD Anderson every 3 months for 2 years or until your disease returns, which ever occurs first. Blood samples (about 4 teaspoons) for gene analysis will be collected within 14 days of completion of chemotherapy, and then every 3 months for 2 years after you enroll in this study. If your colon cancer recurs, a blood sample will be taken at that time also.

You will be asked to fill out the 2 questionnaires described above at the completion of your chemotherapy treatment (if applicable) and 1 and 2 years after your follow-up begins. If your colon cancer recurs, you will be asked to fill out the questionnaires at that time.

If you require surgery for cancer after enrolling in this study, a sample of leftover tissue will be collected for genetic analysis if the surgery is performed at MD Anderson Cancer Center.

You will not be informed of any results of the analysis of your blood and tumor samples or the questionnaires, as this research is exploratory. Your participation in this study will end if your disease returns or 2 years after you begin, whichever occurs first.

This is an investigational study. Taking part in this study requires that you return frequently to MD Anderson. Up to 200 participants will take part in this study. All will be enrolled at MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically proven adenocarcinoma of the colon. Those patients that do not have tissue available at MDACC for analysis will be eligible to participate in the blood, questionnaire and data portion of the study. They will not participate in the tissue portion of this study.
2. AJCC stage II [T3-4(subscript)N0(subscript)M0(subscript)]or stage III [TX(subscript)N1-3(subscript)M0(subscript)].
3. Age >= 14 yrs old.
4. If the patient elects to receive chemotherapy and it is to be administered outside of M. D. Anderson Cancer Center (MDACC), the patient must agree to complete all subsequent surveillance at M.D. Anderson Cancer Center if participating in this clinical trial.
5. Ability to understand and the willingness to sign the written informed consent/authorization document.

Exclusion Criteria:

1. Patients who have initiated adjuvant chemotherapy prior to participating in this study will not be included.
2. Patients with known history of familial adenomatous polyposis (FAP), hereditary nonpolyposis colorectal cancer (HNPCC), and any other hereditary polyposis syndrome (Muir Torre, Gardner's Syndrome, etc) will be excluded since these patients are at increased risk for second primary malignancies and are at higher risk of recurrent disease.
3. No prior malignancies (excluding non-melanomatous skin neoplasms) over the past 5 years.
4. Patients with a known diagnosis of HIV/AIDS or Hepatitis C will be excluded from this study due to their increased risk of second primary malignancies that may complicate appropriate analysis of DFS.
5. Patients who are unable to self-administer the protocol questionnaire will be excluded from this study.

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients 14 years of age and up with colon cancer recently removed by surgery and receiving chemotherapy to try to prevent cancer from returning.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2006-01 (Actual); Primary Completion 2020-01 (Estimated); Study Completion 2020-01 (Estimated)

PRIMARY OUTCOMES:
Occurence of Recurrent Colon Cancer | Information collected at 1, 2 and 3 years after completion of adjuvant chemotherapy or at the time of reoccurrence.
  Study endpoint is occurrence of recurrent colon carcinoma determined radiologically and/or histologically.

CONTACTS AND LOCATIONS:
Overall Officials: Cathy Eng, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org